CLINICAL TRIAL: NCT03939663
Title: Role of Vaginal Misoprostol Prior to IUCD Insertion in Women Who Delivered Only by Elective Caesarean Section.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Enas Mahmoud Mohammed Mohammed Elshahed, MBBCh., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EMMMElshahed
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2018-06

CONDITIONS: IUD Insertion Complication
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo group (Placebo Comparator): 2 tablets vaginally
  Interventions: Drug: Placebo
- misoprostol group (Experimental): 400 mcg vaginally
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — misoprostol 2 tablets
  Other Names: misotac; cytotec
  Arms: misoprostol group
Drug: Placebo — starch pills manufactured to mimic misoprostol 200 mg tablets
  Arms: placebo group

SUMMARY:
Role of vaginal misoprostol prior to IUCD insertion in women who delivered only by elective caesarean section.

DETAILED DESCRIPTION:
Misoprostol ( 400mcg ) vaginally administrated 3 hours prior to IUCD insertion increases the ease and success of insertion and decrease associated pain among women who had delivered only by elective caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* All women will be 20 to 40 years of age.
* Desires IUCD placement and able to participate.
* Negative pregnancy test.
* Willing to follow- up in 6-8 weeks for a standard IUCD follow-up visit.
* Delivered only by cesarean section.

Exclusion Criteria:

* Active cervical infection.
* Current pregnancy.
* Uterine anomaly.
* Fibroid uterus.
* Copper allergy/Wilson's disease.
* Undiagnosed abnormal uterine bleeding.
* Cervical or uterine cancer.
* Allergy to misoprostol.
* Previous vaginal delivery.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
the proportion of failed IUCD insertions regardless of the reason . | during insertion
  pain reported by particiepant during insertion graded from 1 to 10 on visual analogue scale
the degree of difficulty of the IUCD insertion . | during insertion
  Judged as the resistance of the internal cervical os experienced by the investigator and measured by a 5-point scale.

SECONDARY OUTCOMES:
heavy bleeding | 7 days
  heavy bleeding and blood clots
partial or total expulsion | 4 to 6 weeks
  not insitu by U/S

CONTACTS AND LOCATIONS:
Locations (1):
- Enas Mahmoud, Cairo, Egypt